CLINICAL TRIAL: NCT06745557
Title: A Multicentre, Intra-patient Randomised Controlled Phase III Study to Confirm the Efficacy and Safety of DenovoSkin™, a Bilayer Engineered Collagen-based Skin Graft Composed of Autologous Fibroblasts and Keratinocytes, for the Treatment of Patients with Deep Partial and Full-thickness Burns
Brief Title: Phase III Study with an Autologous Dermo-epidermal Skin Substitute for the Treatment of Burns in Adults and Adolescents
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CUTISS AG (Industry)
Collaborators: RCTs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: dS-BA-PIII
Record Dates: First submitted 2024-12-09; First posted 2024-12-20 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Burns
Keywords: Burns; Skin; Scars; Wound healing; Dermis; Epidermis; Thermal burns
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Intervention Model Description: Intra-patient randomisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Option 1 (Other): Location A is the experimental area and Location B is the control area
  Interventions: Biological: denovoSkin(TM); Other: STSG
- Option 2 (Other): Location A is the control area and Location B is the experimental area
  Interventions: Biological: denovoSkin(TM); Other: STSG

INTERVENTIONS:
Biological: denovoSkin(TM) — Transplantation of autologous dermo-epidermal skin substitute denovoSkin(TM) to the experimental area
  Other Names: EHSG-KF
Other: STSG — Transplantation of autologous split-thickness skin to the control area
  Other Names: split-thickness skin graft

SUMMARY:
This multicentre phase III clinical trial will target adults and adolescents of 12 years and older with severe burns to confirm the efficacy and functionality of denovoSkin™ in achieving wound closure and reducing scarring in patients with deep partial and full-thickness burns as compared to split-thickness skin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with deep partial or full-thickness thermal burns of ≥20% total body surface area (TBSA) for which excision and standard of care (SOC) (STSG) are clinically indicated
* Patients of either sex aged ≥12 years
* Signed informed consent from the patient and/or legally authorised representative

Exclusion Criteria:

* Burn wound areas solely located on the head and neck (i.e., test and control areas must NOT be located on head/neck)
* Patients eligible to have all areas autografted in a single surgery or significantly earlier than the end of the manufacturing period of denovoSkin™, for whom the application of denovoSkin™ would delay the standard of care therapies
* Patients with serologic evidence of active hepatitis B virus (HBV) infection (i.e., positive for Hepatitis B surface antigen [HbsAg] or immunoglobulin M total hepatitis B core antibody [anti-HBc]), active hepatitis C infection (hepatitis C virus [HCV] antibody positive), positive human immunodeficiency virus (HIV) serology, or positive Treponema pallidum serology assessed as per local standard of care; cured hepatitis C (defined as documented treatment and negative viral load) is not an exclusion
* Patients with known underlying or concomitant medical conditions that, in the opinion of the Investigator, has the potential to significantly delay wound healing, e.g., glycated haemoglobin (HbA1c) ≥53 mmol/mol and/or systemic skin and connective tissue diseases
* Patients with pre-existing coagulation disorders as defined by international normalised ratio (INR) outside its normal value, a prothrombin time (PT) greater than the upper limit of normal, and fibrinogen less than the lower limit of normal prior to the current hospital admission
* Patients with a history of clinically significant hypersensitivity to amphotericin B, gentamicin, penicillin, streptomycin, or bovine collagen and it's derivatives (e.g. gelatine)
* Previous treatment with denovoSkin™
* Participation in any clinical interventional study within 60 days prior to the first IMP administration in case of monoclonal antibodies and <30 days for all other IMPs
* Patients unwilling or unable to comply with procedures required in this clinical study protocol
* Pregnant or lactating women
* Women of child-bearing potential not using highly effective method(s) of birth control (i.e., with low failure rate <1% per year) throughout the study and/or unwilling to be tested for pregnancy. A negative serum beta-human chorionic gonadotropin (β-hCG) test is required on the day of grafting
* Patient is the Investigator, one of his/her family members, employees, and other dependent persons

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
A composite endpoint whereby success is defined by meeting both of the following criteria: - Wound closure - Scar quality (POSAS v2.0) | 6 months post grafting
  A composite endpoint whereby success is defined by meeting both of the following criteria:
  * Wound closure
  * Scar quality (POSAS v2.0)

SECONDARY OUTCOMES:
Ratio of covered surface area to biopsy site/donor site surface area at 4 weeks post-grafting | 4 weeks
  Ratio of covered surface area to biopsy site/donor site surface area at 4 weeks post-grafting
Assessment of scar contracture | 6 months post grafting
  Assessment of scar contracture
Epithelialisation percentage at 3 months and 6 months post-grafting | 3 months and 6 months post-grafting
  Epithelialisation percentage at 3 months and 6 months post-grafting
Graft take at 14 and 21 days post-grafting | 14 and 21 days post-grafting
  Graft take at 14 and 21 days post-grafting
Assessment of the donor sites | 4 and 10 weeks, and 3, 6, 12, and 24 months post-grafting
  Assessment of the donor sites
Assessment of the grafted burn wounds areas | 4 and 10 weeks and 3, 6, 12, and 24 months post-grafting
  Assessment of the grafted burn wounds areas
Assessment of scar contracture | 12 and 24 months post-grafting
  Assessment of scar contracture

OTHER OUTCOMES:
Assessment of safety and tolerability using the National Cancer Institute-CTCAE v5.0 throughout the study: - Assessment of the incidence of treatment-emergent adverse events (TEAEs), total AEs, and serious adverse events (SAEs) | 24 months
  Assessment of safety and tolerability using the National Cancer Institute-CTCAE v5.0 throughout the study:
  - Assessment of the incidence of treatment-emergent adverse events (TEAEs), total AEs, and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Rode Kruis Ziekenhuis, Beverwijk, Netherlands

IPD SHARING:
Plan to Share IPD: No